CLINICAL TRIAL: NCT02277171
Title: Prospective, Phase I, Single-Center, Evaluation of the Safety and Tolerability of Nitric Oxide Impregnated Urinary Catheters in Patients Undergoing Radical Prostatectomy
Brief Title: Evaluation of Safety and Tolerability of Nitric Oxide Impregnated Urinary Catheters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enox Israel Ltd (Industry)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ENOX PHASE I_1.1
Record Dates: First submitted 2014-10-19; First posted 2014-10-28 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Urinary Tract Infection; Bacteriuria
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitric oxide impregnated catheter (Experimental)
  Interventions: Device: Nitric Oxide impregnated catheter

INTERVENTIONS:
Device: Nitric Oxide impregnated catheter — Patients undergoing radical prostatectomy will be catheterized for 7-14 days with Nitric Oxide impregnated Foley catheters

SUMMARY:
According to the World Health Organization, hundreds of millions of patients are affected by health-care associated infections worldwide each year, resulting in prolonged hospital stays, long-term disabilities, deaths, and financial losses for health systems. The most common hospital-acquired infection is Urinary Tract Infection (UTI), accounting for almost 40% of all nosocomial infections. Most hospital-acquired UTIs are associated with catheterization. In fact, urinary catheter-related bacteriuria is the most common health care associated infection worldwide. Catheter-associated UTI (CAUTI) develops following adhesion of planktonic bacteria to the surface of the catheter and colonization, creating a persistent environment called a biofilm. The nature of biofilm structure together with the physiological attributes of biofilm organisms confers an inherent resistance to various antimicrobial agents such as antibiotics, disinfectants or germicides, augmenting the potential of these pathogens to cause infections in catheterized patients.

Nitric oxide (NO) is a naturally-produced gas molecule with broad-spectrum antimicrobial activity. NO is used in the clinics to treat pulmonary hypertension in neonates and adults. Studies have shown that low-dose NO is associated with prevention of biofilm formation, biofilm dispersal and elimination of bacteria. It is suggested that NO prevents bacteria attachment to catheter surfaces and inhibits biofilm formation in a mechanism involving reduction and modification of proteins that mediate cell-substrate and cell-cell interactions.

The investigators team, using a proprietary technology impregnate urinary catheters with NO (i.e. NO-impregnated catheters). These catheters release low concentration of NO following exposure to urine over a 14-day period. In vitro studies showed that NO-impregnated catheters prevent bacterial colonization and biofilm formation of Escherichia coli on exterior and luminal surfaces of the catheters. In addition, NO released from these catheters is able to eradicate up to 4log colony forming unit/ml of bacteria within the surrounding media. Moreover, NO-impregnated catheters exhibit superior performance compared to silver-coated catheters, and similar anti-infective properties compared to antibiotic-coated catheters.

Primary objectives: To assess the safety and tolerability of NO-impregnated catheters in patients older than 18 years old undergoing radical prostatectomy and catheterized for 7-14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients before radical prostatectomy at the Department of Urology in Beilinson Medical Center, which will be catheterized for 7-14 days.
2. Age: ≥ 18 years.
3. Patients with a life expectancy of more than 12 months.
4. The investigator has completed a medical history and a physical examination to assure that the patients meets all study enrollment criteria.
5. The patient is willing and able to read, understand and sign the study specific informed consent form.

Exclusion Criteria:

1. A urinary culture demonstrating UTI before surgery.
2. A patient with an indwelling urinary catheter prior to surgery.
3. Expected life expectancy of less than 12 months.
4. Concurrent illness, disability or geographical residence that would hamper study participation.
5. Patients with underlying diseases such as heart disease, lung disease, skin disease or infection involving the penis, scrotum and groin, immunocompromised patients (transplant recipients, HIV carriers) or any other disease or condition that according to the physician opinion will influence the study results.
6. Patients with known urethral stricture.
7. Patients with recurrent UTIs.
8. Current participation in another clinical investigation of a medical device or a drug or has participated in such a study within 30 days prior to study enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events associated with Nitric Oxide impregnated catheters | 30-45 days
Proportion of patients (%) who prematurely discontinued the study due to adverse events or severe adverse events associated with Nitric oxide impregnated catheters | 30-45 days

SECONDARY OUTCOMES:
Measuring biofilm forming bacteria on the surface of Nitric Oxide impregnated and non impregnated Foley catheters after indwelling for 7 to 14 days | 7-14 days
Measuring bacteriuria (by urine culture) for Nitric Oxide impregnated and non impregnated Foley catheters prior to insertion, 1 day after insertion, every day during hospitalization, on catheter removal day, and 30 days after catheterization | 30-45 days
Measuring number of urinary tract infection (UTI) events following catheterization with Nitric Oxide impregnated and non impregnated Foley catheters | 30-45 days
Proportion of patients (%) who prematurely discontinued the study for any reason | 30-45 days

CONTACTS AND LOCATIONS:
Overall Officials: David Greenberg, prof., Study Chair — ENOX

REFERENCES:
- [Background] Regev-Shoshani G, Ko M, Miller C, Av-Gay Y. Slow release of nitric oxide from charged catheters and its effect on biofilm formation by Escherichia coli. Antimicrob Agents Chemother. 2010 Jan;54(1):273-9. doi: 10.1128/AAC.00511-09. Epub 2009 Nov 2. PMID 19884372
- [Background] Regev-Shoshani G, Ko M, Crowe A, Av-Gay Y. Comparative efficacy of commercially available and emerging antimicrobial urinary catheters against bacteriuria caused by E. coli in vitro. Urology. 2011 Aug;78(2):334-9. doi: 10.1016/j.urology.2011.02.063. PMID 21820571
- [Background] Barraud N, Storey MV, Moore ZP, Webb JS, Rice SA, Kjelleberg S. Nitric oxide-mediated dispersal in single- and multi-species biofilms of clinically and industrially relevant microorganisms. Microb Biotechnol. 2009 May;2(3):370-8. doi: 10.1111/j.1751-7915.2009.00098.x. Epub 2009 Mar 13. PMID 21261931
- [Background] Charville GW, Hetrick EM, Geer CB, Schoenfisch MH. Reduced bacterial adhesion to fibrinogen-coated substrates via nitric oxide release. Biomaterials. 2008 Oct;29(30):4039-44. doi: 10.1016/j.biomaterials.2008.07.005. Epub 2008 Jul 26. PMID 18657857
- [Background] Ramritu P, Halton K, Collignon P, Cook D, Fraenkel D, Battistutta D, Whitby M, Graves N. A systematic review comparing the relative effectiveness of antimicrobial-coated catheters in intensive care units. Am J Infect Control. 2008 Mar;36(2):104-17. doi: 10.1016/j.ajic.2007.02.012. PMID 18313512
- [Background] Siddiq DM, Darouiche RO. New strategies to prevent catheter-associated urinary tract infections. Nat Rev Urol. 2012 Apr 17;9(6):305-14. doi: 10.1038/nrurol.2012.68. PMID 22508462
- [Background] Parida S, Mishra SK. Urinary tract infections in the critical care unit: A brief review. Indian J Crit Care Med. 2013 Nov;17(6):370-4. doi: 10.4103/0972-5229.123451. PMID 24501490